CLINICAL TRIAL: NCT04232709
Title: Evaluating the CAREchart@Home™ Program for Enhancing After-hours Care of Cancer Patients in Ontario: A Pilot Randomized Controlled Trial
Brief Title: Evaluating the CAREchart@Home™ Program for Enhancing After-hours Cancer Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to unforeseen circumstances, the funder decided to discontinue all funding.
Sponsor: Women's College Hospital (Other)
Collaborators: Southlake Regional Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: WCHCCH-001
Record Dates: First submitted 2019-03-04; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Cancer
Keywords: systemic therapy; chemotherapy; targeted therapy; immunotherapy; after-hours telemedicine; shared electronic patient record; symptom management; oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- After-hours care (No Intervention): Patients in the after-hours care (AH) group will receive the usual (telemedicine) care. That is, they will have the option to call the after-hours centre and receive help from the oncology nurses using the COSTaRS practice guides to manage their after-hours symptoms.
- After-hours care w/personal health info (Experimental): Patients in the after-hours care with personal health information (AH-PHI) group will also receive the usual (telemedicine) care. However, if they call the telemedicine service, the oncology nurses will have access to some of their personal health information from the cancer centre (i.e., a shared electronic patient record) via the MedChart platform.
  Interventions: Other: Shared electronic patient record

INTERVENTIONS:
Other: Shared electronic patient record — MedChart allows access to a shared electronic patient record that contains selected information related to a patient's cancer treatment. If a patient contacts the after-hours telemedicine service, the oncology nurse will have access to this shared record
  Other Names: MedChart
  Arms: After-hours care w/personal health info

SUMMARY:
The objective of the current project is to pilot the evaluation of the health and economic benefits of having online access to health information in the context of providing telemedicine support for oncology patients receiving outpatient systemic therapy in Ontario. This pilot study will determine the feasibility of conducting a full-scale randomized controlled trial that could definitively determine whether the addition of access to patients' health information in the after-hours telemedicine program reduces emergency department use, affect patients' experience of care, or improve patient-reported health.

The study will be conducted at, and with patients from, the Stronach Regional Cancer Centre (SRCC) at Southlake. Eligible patients will be adults (at least 18 years of age) with a confirmed cancer diagnosis, and initiating or continuing treatment with systemic therapy at the SRCC. Prospective patients will be randomized across two arms. Recruitment will take place during a 6.5-month recruitment period and followed up for a period of 3 months.

DETAILED DESCRIPTION:
Advances in systemic therapy (including oral or intravenously injected anti-cancer drugs) have led to the improvement in overall survival for many cancers and more than half of patients diagnosed with cancer will receive some form of systemic therapy. Unfortunately, Cancer Care Ontario (CCO) data indicates that up to 50% of patients will experience treatment-related side effects resulting in a visit to the emergency department (ED) or admission to hospital within 4 weeks of receiving chemotherapy - the most common form of systemic therapy. Despite differences in international healthcare systems, it is useful to note that one US-based study found that approximately 25% of total ED costs during cancer treatment could be potentially preventable, presenting a significant opportunity to lower health system costs related to cancer care.

While most systemic therapy is delivered in cancer clinics which operate during business hours, data shows that a significant portion of unplanned ED visits and hospital admissions occur after-hours, that is, on evenings and weekends. One of the strategic priorities of CCO's 2014-2019 Systemic Treatment Provincial Plan was to reduce ED utilization through enhanced management of toxicity due to treatment with one avenue being the provision of symptom management services through alternate models of care, especially during after-hour time periods.

In July 2016, Bayshore Healthcare Ltd. introduced a program to provide after-hours symptom management support for oncology patients receiving systemic therapy. The program runs Monday to Friday 6:00pm - 8:30am, and Saturday 8:30am to Monday 8:30am, including statutory holidays and involves highly trained oncology nursing staff answering telephone calls from patients related to symptom management. In two separate partnerships in 2016, Southlake Regional Health Centre partnered with Bayshore HealthCare Ltd. to pilot the after-hours telephone symptom management program and also initiated a concurrent, but completely separate pilot with MedChart Inc. to offer Southlake patients (and their circle of care) online access to medical records, primarily outside the cancer program. MedChart's technology is a cloud-based, online Consumer Moderated Health Information Exchange (CME) network that connects to healthcare providers and provides access to health records in any format.

While at least one study has reported a reduction in ED visits, over four years, after the introduction of telephone support with physician access to medical records, the causal pathway connecting the provision of the medical records with reduced ED visits and health system costs is largely unexplored. As such, it is unclear whether there are outcomes, other than ED utilization, that may also be scientifically interesting and/or more feasible to capture. Furthermore, there are no recent studies that prospectively compared the provision of after-hours services with and without medical records.

The objective of the current project is to pilot the evaluation of the health and economic benefits of having online access to health information in the context of providing telemedicine support for oncology patients receiving outpatient systemic therapy in Ontario. This pilot study will determine the feasibility of conducting a full-scale randomized controlled trial (RCT) that could definitively determine whether the addition of access to patients' health information in the after-hours telemedicine program reduces emergency department use, affects patients' experience of care, or improves patient-reported health. The evaluation will focus on the shared electronic patient record (provided by MedChart) in the context of Bayshore's after-hours telemedicine program (CAREchart@home).

This will be a single-centre, non-blinded, two-arm pilot RCT. Once recruited, patients will be randomized to one of two study arms: (1) the control arm, which constitutes usual care - access to after-hours telemedicine (AH); and (2) the intervention arm - access to after-hours telemedicine with some cancer-related personal health information (AH-PHI), i.e. CAREchart@home™. Recruitment will take place during a 6.5-month recruitment time period and all patients will be followed up for a period of 3 months during which patients will complete a series of questionnaires and data from institutional records will be compiled.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cancer diagnosis (all cancers, all stages)
* Initiating or continuing treatment with systemic therapy (oral or injected/IV; excluding hormonal therapy for breast or prostate cancer) at Stronach Regional Cancer Centre at Southlake

Exclusion Criteria:

* Being treated with radiation
* Unable to read or understand spoken English (Required for completing the questionnaires)
* Unable to utilize the after-hours services due to cognitive impairment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients willing to be randomized | 9.5 Months
  The proportion of patients willing to be randomized
Proportion of enrolled patients lost to follow up | 9.5 Months
  The proportion of enrolled patients lost to follow up in each randomized group
Number of attempted questionnaires relative to number of questionnaires that should have been completed | 9.5 Months
  The number of completed questionnaires for both patient participants and healthcare provider participants in relation to the total number of times a questionnaire should have been completed
Number of completed questionnaires relative to number of questionnaires that should have been completed | 9.5 Months
  The number of attempted questionnaires for both patient participants and healthcare provider participants in relation to the total number of times a questionnaire should have been completed
Percent of total emergency department (ED) visits reported that occurred at Southlake | 9.5 Months
  Comparison of total self-reported ED visits to total ED visits recorded in institutional records
Time to complete questionnaire battery | 9.5 Months
  Estimation of time required for patients to complete the questionnaires at each timepoint
Completion rate for satisfaction survey | 9.5 Months
  Percent of callers for whom Bayshore's satisfaction survey results were obtained

SECONDARY OUTCOMES:
Self-reported health service utilization | 3 Months
  Total number of encounters with the health system for any concern, including cancer-related symptom management.
Hospital-reported health service utilization: Emergency Department Visits | 3 Months
  The total number of emergency department visits
Hospital-reported health service utilization: Outcomes of ED Visits | 3 Months
  The outcomes of the emergency department visits
Hospital-reported health service utilization: Length of Hospital Stay | 3 Months
  The total length of stay for any admission to the hospital
Edmonton Symptom Assessment System-revised (ESAS-r) Scale | 3 Months
  Self-reported measurement of the severity of nine common symptoms of cancer, at the time of questionnaire completion
Functional Assessment of Cancer Therapy - General (FACT-G) Scale | 3 Months
  Patient-reported assessment of health-related quality of life, over the past week, for patients undergoing cancer therapy
Prompt Access to Care (PAC) Scale | 3 Months
  Measurement of a cancer patient's perception of their ability to reach or see an oncology professional, as required, at various times of the day and on different days of the week
Continuity of Care (CoC) Scale | 3 Months
  Measurement of a cancer patient's perception of continuity of care across all healthcare professionals in the cancer care continuum
Prevented health service utilization | 3 Months
  Frequency of reports of a health service that a patient would have accessed if they did not have access to the after-hours service
Efficiency of after-hours service advice | 3 Months
  Proportion of calls that were handled by telephone advice alone, that is, those calls that were not followed by any unplanned referrals or visits to other healthcare professional within 2 weeks of the after-hours service encounter
Patient confidence | 3 Months
  Patients' level of confidence in the advice they received through the after-hours service
Perceived reliability of the after-hours service encounter | 3 Months
  Patients' perceived reliability of the after-hours service encounter which will be measured as agreement with a statement regarding the similarity of the encounter to an in-person visit
Provider confidence (measured using a modified version of the C-scale) | 3 Months
  Assessment of a nurse's confidence in relation to various aspects of the triage encounter

CONTACTS AND LOCATIONS:
Overall Officials: Sacha Bhatia, MD, FRCPC, MBA, Principal Investigator — Women's College Hospital; Peter Anglin, MD, FRCPC, MBA, Principal Investigator — Southlake Regional Health Centre
Locations (1):
- Southlake Regional Health Centre, Newmarket, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barbera L, Atzema C, Sutradhar R, Seow H, Howell D, Husain A, Sussman J, Earle C, Liu Y, Dudgeon D. Do patient-reported symptoms predict emergency department visits in cancer patients? A population-based analysis. Ann Emerg Med. 2013 Apr;61(4):427-437.e5. doi: 10.1016/j.annemergmed.2012.10.010. Epub 2013 Jan 4. PMID 23290526
- [Background] Cancer Care Ontario. (2014). Quality Person-Centred Systemic Treatment in Ontario, 2014-2019 (pp. 1-46). Toronto, ON: Cancer Care Ontario.
- [Background] Cancer Quality Council of Ontario. (2016, October). Cancer Safety Quality Index: Unplanned Hospital Visits During Chemotherapy. Retrieved March 23, 2018, from http://www.csqi.on.ca/by_patient_journey/treatment/unplanned_hospital_visits_during_chemotherapy/
- [Background] Ferrer-Roca O, Subirana R. A four-year study of telephone support for oncology patients using a non-supervised call centre. J Telemed Telecare. 2002;8(6):331-6. doi: 10.1258/135763302320939211. PMID 12537920
- [Background] Kurtz ME, Kurtz JC, Given CW, Given B. Effects of a symptom control intervention on utilization of health care services among cancer patients. Med Sci Monit. 2006 Jul;12(7):CR319-24. Epub 2006 Jun 28. PMID 16810138
- [Background] Palumbo MO, Kavan P, Miller WH Jr, Panasci L, Assouline S, Johnson N, Cohen V, Patenaude F, Pollak M, Jagoe RT, Batist G. Systemic cancer therapy: achievements and challenges that lie ahead. Front Pharmacol. 2013 May 7;4:57. doi: 10.3389/fphar.2013.00057. eCollection 2013. PMID 23675348
- [Background] Panattoni, L., Fedorenko, C. R., Kreizenbeck, K. L., Greenlee, S., Walker, J. R., Greenwood-Hickman, M. A., et al. (2017). Costs of potentially preventable emergency department use during cancer treatment: A regional study [Abstract]. Journal of Clinical Oncology / 2017 ASCO Annual Meeting, 35(8_suppl), Abst 6505. http://doi.org/10.1200/JCO.2017.35.8_suppl.2